CLINICAL TRIAL: NCT01026935
Title: The Effect of Mesh Type on Pain After Surgery for Inguinal Hernia. Randomized Clinical Trial of Lichtenstein Operation With Sutured Polypropylene Patch or Self-adhesive ProGrip Patch.
Brief Title: The Outcome After Lichtenstein Operation vs. ProGrip Patch Repair of Inguinal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Jaana Vironen, MD PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 231268
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2009-12

CONDITIONS: Inguinal Hernia; Primary; Unilateral
Keywords: open mesh repair; sutured; non-sutured; pro-grip; postoperative pain
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sutured mesh (Experimental): 200 patients are randomized to inguinal hernia repair with sutured light weight (38g/m2) polypropylene mesh (Lichtenstein repair)
  Interventions: Device: Open inguinal hernia repair
- non-sutured mesh (Experimental): 200 patients are randomized to receive a light weight mesh that adheres to tissues with polylactic micro hooks without sutures
  Interventions: Device: Open inguinal hernia repair

INTERVENTIONS:
Device: Open inguinal hernia repair — Altogether 400 patients are randomized to receive an open mesh repair with either sutured light weight mesh (38g/m2) or with a non-sutured light weight polypropylene mesh that adheres to tissues with polylactic micro hooks
  Other Names: Parietene Light; Parietene ProGrip

SUMMARY:
For the present study, 400 consecutive men with unilateral primary inguinal hernia are randomized to Lichtenstein repair using either light weight polypropylene mesh (38g/m2) or light weight ProGrip mesh. ProGrip mesh adheres to tissues with polylactic micro hooks without suturing. The primary aim is to examine, whether the ProGrip mesh produces less pain than sutured polypropylene mesh. Secondary outcomes are operation time and convalescence as well as recurrence rate. ProGrip mesh is supposed to be faster to apply as no sutures are needed, which may compensate for its higher cost. The patients are blinded to which mesh they receive.

ELIGIBILITY:
Inclusion Criteria:

* primary unilateral inguinal hernia

Exclusion Criteria:

* not willing to participate
* not capable to understand or fill in the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2008-02; Primary Completion 2010-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
postoperative complaints | One year

SECONDARY OUTCOMES:
Recurrence rate | One year

CONTACTS AND LOCATIONS:
Overall Officials: Jaana Vironen, MD PhD, Principal Investigator — HUCH Jorvi Hospital
Locations (2):
- Finland (2):
  - HUCH Jorvi Hospital, department of Surgery, Espoo
  - HUCH Surgical Hospital, Dept of Surgery, Helsinki

REFERENCES:
- [Derived] Pierides G, Scheinin T, Remes V, Hermunen K, Vironen J. Randomized comparison of self-fixating and sutured mesh in open inguinal hernia repair. Br J Surg. 2012 May;99(5):630-6. doi: 10.1002/bjs.8705. Epub 2012 Feb 23. PMID 22362035